CLINICAL TRIAL: NCT01413737
Title: Postoperative Results of Surgical Treatment of Lung Cancer After 30 Days
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 4.2005.1826
Record Dates: First submitted 2005-09-22; First posted 2011-08-10 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a retrospective, descriptive analysis of (1) 30 day postoperative results of surgery for lung cancer, (2) 30 day outcome predictors - compared to an earlier similar study in the same hospital (St Olav University Hospital, Trondheim, Norway).

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer patients after surgery in 2002-2004 at dept for Heart and Lung Surgery, St.Olavs University Hospital, Trondheim, Norway.

Exclusion Criteria:

* Carcinoid tumor, small-cell lung cancer, lung metastases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: lung cancer patients after surgery at St Olavs University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rune Haaverstad, Ph.D, Study Chair — National Taiwan Normal University
Locations (2):
- Norway (2):
  - NTNU, Trondheim, Sør-Trøndelag
  - NTNU, Trondheim

REFERENCES:
- [Result] Hjelde H, Sundstrom S, Odegard A, Hatlinghus S, Abusland AB, Haaverstad R. [Recurrence and survival after surgical treatment of lung cancer]. Tidsskr Nor Laegeforen. 2010 Jan 14;130(1):25-8. doi: 10.4045/tidsskr.09.0689. Norwegian. PMID 20094119
- [Result] Roth K, Nilsen TI, Hatlen E, Sorensen KS, Hole T, Haaverstad R. Predictors of long time survival after lung cancer surgery: a retrospective cohort study. BMC Pulm Med. 2008 Oct 27;8:22. doi: 10.1186/1471-2466-8-22. PMID 18954454